CLINICAL TRIAL: NCT03716765
Title: Locally Injected Vitamin D as a Non-surgical Modality for Periodontal Regeneration of Infrabony Defects: Prospective Study
Brief Title: Locally Injected Vit D as a Non-surgical Modality for Periodontal Regeneration of Infrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, nermin mohammed ahmed yussif, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1236
Record Dates: First submitted 2018-10-13; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Periodontal Bone Loss; Periodontal Pocket
MeSH Terms: conditions — Alveolar Bone Loss; Periodontal Pocket

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- non-surgical periodontal regeneration (Experimental): non-surgical periodontal regeneration using locally injected vitamin d to treat the infrabony defect
  Interventions: Dietary Supplement: locally injected vitamin D
- surgical peridoontal regeneration (Active Comparator): surgical periodontal regeneration using bone graft and collagen barrier
  Interventions: Dietary Supplement: locally injected vitamin D

INTERVENTIONS:
Dietary Supplement: locally injected vitamin D — locally injected vitamin d as non surgical method for periodontal regeneration of vertical bony defects
  Other Names: non-surgical periodontal rgeneration

SUMMARY:
vitamin D has great role in bone regenration and soft tissue health. in the past periodontal regeneration was performed using bone graft and barrier membrane

DETAILED DESCRIPTION:
there was no previous studies used the locally injected vitamin d in periodontal regeneration. therefore, we intended to study the effect of locally injected vitamin D in peridoontal regerneration in comparison with the conventional surgical technique

ELIGIBILITY:
Inclusion Criteria:

* patients with infrabony vertical defects
* systemically free patients
* periodontally affected patients

Exclusion Criteria:

* patients with systemic diseases
* smokers
* pregnency

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
radiographic interproximal bone level | 6 months
  radiographic interproximal bone level

CONTACTS AND LOCATIONS:
Overall Officials: nermin yussif, Study Director — Modern Science and Arts University

IPD SHARING:
Plan to Share IPD: No